CLINICAL TRIAL: NCT00228956
Title: A Multi-Center Randomized Clinical Trial Correlating the Effects of 24 Months of Exemestane or Letrozole on Surrogate Markers of Response With Aromatase Polymorphism
Brief Title: Aromatase Inhibitor Clinical Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Collaborators: Indiana University School of Medicine (Other); Office of Research on Women's Health (ORWH) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 0412-14; U01GM061373-06 (NIH); NCT00263913 (obsolete NCT alias)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2005-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Aromatase Inhibitor; Letrozole; Exemestane
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum and Plasma Urine

INTERVENTIONS:
Drug: pharmacodynamic analysis — Exemestane 25mg po daily or Letrozole 2.5mg po daily

SUMMARY:
You are invited to participate in a research study looking at metabolism (breakdown) and effects of aromatase inhibitors. The purpose of this research is to try to identify which women who take an aromatase inhibitor are more likely to have certain benefits or side effects from the drug. We will do so by determining whether there are differences that normally occur in genes that you have inherited from your parents that might influence the way individuals respond to medications. If you agree to participate in this study, you will be asked to sign this informed consent form.

DETAILED DESCRIPTION:
Primary Objective To determine baseline breast density and the change in this parameter that occurs in post-menopausal women with hormone-receptor positive primary breast cancer taking letrozole or exemestane for 24 months, and to correlate the changes with wild type or variant aromatase (CYP19).

Secondary Objectives

1. To determine serum estrone sulfate concentrations at baseline and following one, three and 24 months of letrozole or exemestane therapy. We will use these concentrations to test the hypothesis that candidate genes involved in estrogen metabolism in post-menopausal women, or in the metabolism and disposition of exemestane or letrozole, influence the ability of aromatase inhibitors to reduce estrogen metabolite concentrations.
2. To determine bone density and bone turnover metabolites in post-menopausal women. The bone densitometry will be done at baseline and following 24 months of letrozole or exemestane therapy. The bone turnover metabolites will be done at baseline, three, six and 24 months following letrozole or exemestane therapy. These data will allow us to test the hypothesis that variants in candidate genes involved in estrogen metabolism or signaling alter the ability of exemestane or letrozole to bring about changes in bone.
3. To objectively measure hot flashes at baseline and monitor changes in hot flashes after one, three, six and 12 months of letrozole or exemestane therapy, and correlate these changes with serum FSH and LH concentrations. We will test the hypothesis that aromatase or estrogen receptor variants influence the phenotype of hot flashes at baseline or during treatment as part of a broader approach in which we will test for associations with other candidate genes involved in estrogen metabolism and signaling, or with aromatase inhibitor metabolism and disposition.
4. To measure changes in symptoms that may be related to hot flashes and estrogen deprivation such as menopausal symptoms, mood (depression, anxiety), sleep quality and sleep disturbance and overall quality of life at baseline and after one, three, six, twelve and 24 months of treatment.
5. To measure changes in fasting lipid profiles at baseline and after 3 months of letrozole or exemestane therapy.
6. To determine letrozole and exemestane serum concentrations at baseline and after one, three, six, twelve and 24 months of treatment to test the hypothesis that genetic variants in drug metabolizing enzymes predict drug concentrations and effects.
7. To measure serum thyroid binding globulin and sex hormone binding globulin concentrations before and after one and three months of treatment, to test whether changes in these parameters brought about by aromatase inhibitor treatment are altered by genetic variants in candidate genes involved in estrogen metabolism or signaling.
8. To categorize the rheumatic adverse effects experienced by patients on aromatase inhibitors by specifically characterizing anatomic structures involved and documenting the presence or absence of inflammation in these tissues; to identify any correlations between changes in musculoskeletal symptoms and the duration of therapy with aromatase inhibitors; and to identify any correlations between changes in musculoskeletal symptoms and levels of circulating estrogen and its metabolites. This will be done at baseline and after one, three, six, twelve and 24 months of treatment.
9. To determine a number of specific platelet functions before and after 3 months of letrozole and exemestane treatment. This is a sub-study that will be performed only at the Indiana University site. Platelet function will be measured by ex vivo platelet aggregation tests. Production of regulators of platelet function, including thromboxane A2 (TXA2), proscyclin (PGI2) and serotonin will also be assessed. These data will allow us to test the hypothesis that genetic polymorphisms in candidate genes in estrogen-regulated pathways alter the effect of letrozole and exemestane treatment on platelet activity, which may be relevant to their effects on cardiac risks.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender.
2. Post-menopausal status, defined as:

   * age > 60; or
   * less than age 60 and the last menstrual period >12 months prior to enrollment in trial if intact uterus/ovaries; or,
   * less than age 60 and the last menstrual period 6-12 months prior to enrollment in trial if intact uterus/ovaries and meets biochemical criteria for menopause (FSH and estradiol levels within institutional standards for menopausal status) NOTE: These subjects will have serum estradiol levels checked at visits 0, 1, 3, 6 and 12 months to check for continued menopausal status; or,
   * less than age 60 and history of bilateral oophorectomy; or,
   * less than age 60 and has a history of hysterectomy and meets biochemical criteria for menopause (FSH and estradiol levels within institutional standards for menopausal status).

   NOTE: These subjects will have serum estradiol levels checked at visits 0, 1, 3, 6 and 12 months to check for continued menopausal status; or,
   * less than age 60 and taking medication designed to suppress ovarian function and meets biochemical criteria for menopause (estradiol levels within institutional standards for menopausal status). Women would have had to be taking the drug for at least 30 days prior to entering the study.

   NOTE: While the patient is being treated with a GnRh agonist (luprolide or goserelin), serum estradiol levels will be checked at visits 0, 1, 3, 6 and 12 months to check for menopausal status.
3. Patients with histologically proven ductal carcinoma in situ (DCIS/stage 0) or stage I-III invasive carcinoma of the breast that is ER and/or PR positive by immunohistochemical staining, who are considering aromatase inhibitor therapy. Patients must have completed any adjuvant chemotherapy. Patients may have received preoperative chemotherapy. Patients should have also completed local therapy; however, enrollment/initiation of aromatase inhibitor on study may be done prior to completion of radiation therapy. Women may receive the aromatase inhibitor on this study as initial adjuvant hormonal treatment or following adjuvant tamoxifen.
4. ECOG performance status 0-2.
5. The patient is aware of the nature of her diagnosis, understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

1. History of bilateral mastectomy.
2. History of radiation to the contralateral breast.
3. Prior use of an aromatase inhibitor.
4. Personal history of the following cancers: ovarian, endometrial, fallopian tube and primary peritoneal carcinomatosis.
5. Presence of implant in contra-lateral breast.
6. Women with history of breast reduction should be entered at the discretion of the investigator. Breast reduction during the two years of the trial is strongly discouraged.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2005-01; Study Completion 2009-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Storniolo, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - UMCCC, Ann Arbor, Michigan

REFERENCES:
- [Derived] Kidwell KM, Harte SE, Hayes DF, Storniolo AM, Carpenter J, Flockhart DA, Stearns V, Clauw DJ, Williams DA, Henry NL. Patient-reported symptoms and discontinuation of adjuvant aromatase inhibitor therapy. Cancer. 2014 Aug 15;120(16):2403-11. doi: 10.1002/cncr.28756. Epub 2014 May 6. PMID 24802413
- [Derived] Henry NL, Pchejetski D, A'Hern R, Nguyen AT, Charles P, Waxman J, Li L, Storniolo AM, Hayes DF, Flockhart DA, Stearns V, Stebbing J. Inflammatory cytokines and aromatase inhibitor-associated musculoskeletal syndrome: a case-control study. Br J Cancer. 2010 Jul 27;103(3):291-6. doi: 10.1038/sj.bjc.6605768. Epub 2010 Jul 6. PMID 20606683
- [Derived] Henry NL, Jacobson JA, Banerjee M, Hayden J, Smerage JB, Van Poznak C, Storniolo AM, Stearns V, Hayes DF. A prospective study of aromatase inhibitor-associated musculoskeletal symptoms and abnormalities on serial high-resolution wrist ultrasonography. Cancer. 2010 Sep 15;116(18):4360-7. doi: 10.1002/cncr.25385. PMID 20549827
- [Derived] Bao T, Fetting J, Mumford L, Zorzi J, Shahverdi K, Jeter S, Herlong F, Stearns V, Lee L. Severe prolonged cholestatic hepatitis caused by exemestane. Breast Cancer Res Treat. 2010 Jun;121(3):789-91. doi: 10.1007/s10549-009-0576-x. Epub 2009 Oct 16. No abstract available. PMID 19834799
- See also: The Pharmacogenetics and Pharmacogenomics Knowledge Base — http://www.pharmgkb.org